CLINICAL TRIAL: NCT06287879
Title: Function and Morphological Characteristics of Meibomian Gland in Patients With Renal Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20231121
Record Dates: First submitted 2024-02-01; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye; MGD-Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Subjects were treated with Roxadustat for renal anemia
  Interventions: Diagnostic Test: Dry eye examination
- EPO (Active Comparator): Subjects were treated with EPO for renal anemia
  Interventions: Diagnostic Test: Dry eye examination

INTERVENTIONS:
Diagnostic Test: Dry eye examination — 1. Lacrimal river height
  2. tear break-up time
  3. tear-film lipid layer thickness
  4. meibomian glands two-dimensional digital infrared images

SUMMARY:
Renal anemia refers to anemia in which the absolute or relative production of erythropoietin (EPO) is insufficient due to various kidney diseases, and uremic toxins affect erythropoietin production and its lifespan. Common treatment drugs for renal anemia include erythropoietin EPO and Roxadustat (FG-4592).

Medical history information was collected from patients with renal anemia who visited the ophthalmology department with dry eye symptoms.

This study will help to determine the function and morphological characteristics of meibomian gland in patients with renal anemia

DETAILED DESCRIPTION:
1. Collect medical records of patients with renal anemia who visited the ophthalmology outpatient department of Zhongnan Hospital and hospitalized patients with renal anemia
2. Patients were divided into Rosallistat group, and EPO group according to their drug use history.
3. The dry eye analysis results of all patients were collected, and the lacrimal river height, tear film rupture time and meibomian gland grade were counted. The results of dry eye examination were analyzed statistically.
4. Complete data collection, conduct statistical analysis, and evaluate the analysis results.

ELIGIBILITY:
Inclusion Criteria:

* long-term use of Roxadustat or erythropoietin for renal anemia

Exclusion Criteria:

* contact lens wearer, history of eye surgeries, systemic health conditions affecting ocular health and those who were unable to cooperate with examinations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Lacrimal river height | Immediately and six months later
  Measured by dry eye analyzer machine
tear break-up time | Immediately and six months later
  Measured by dry eye analyzer machine
tear-film lipid layer thickness | Immediately and six months later
  Measured by dry eye analyzer machine
meibomian glands two-dimensional digital infrared images | Immediately and six months later
  Measured by dry eye analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China